CLINICAL TRIAL: NCT01019798
Title: Phase II Study of Salvage Therapy With Sunitinib,Docetaxel and Platinum on Metastatic or Unresectable Non Small Cell Lung Cancer
Brief Title: Salvage Therapy With Sunitinib,Docetaxel and Platinum on Metastatic or Unresectable Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: Pfizer (Industry); TTY Biopharm (Industry)
Responsible Party: Cheng-Jeng Tai, M.D., Director, Hematology-Oncology, Department of Medicine., Taipei Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-01-08-03
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; sunitinib; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sunitinib; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label (Experimental)
  Interventions: Drug: sunitinib, docetaxel, cisplatin

INTERVENTIONS:
Drug: sunitinib, docetaxel, cisplatin — 1. Sunitinib given 10 days within 14 days of each cycle。
  2. Sunitinib 25 mg/day with adjust dosage according to patient's condition, but should return to 25 mg when feasible or should withdraw from this study.
  3. Docetaxel 40-50 mg/m2, cisplatin 50 mg/m2 every 2 weeks.
  4. Overall 12 cycles (24 weeks)
  Other Names: docetaxel(tyxant)

SUMMARY:
Sunitinib shows anti-tumor activity in a variety of human non-small cell lung tumor ex vivo models. Many Phases II and III clinical trials of sunitinib in several solid tumors are completed or still ongoing. So far, the efficacy of sunitinb has been confirmed by the phase III trial for imatinib-resistance or intolerance advanced gastrointestinal stromal tumor patients. And sutent was approved to effective by two phase II trials in advanced renal cell carcinoma patients after failure of immunotherapies, and one phase III trial in treatment-naive advanced renal carcinoma patients. Sunitinib (SUTENT ®) has been approved by U.S. Food and Drug Administration (FDA) for the treatment of advanced renal carcinoma patients and in gastrointestinal stromal tumor patients who are intolerant or progressed after imatinib mesylate. European Medicines Agency (EMEA) conditionally granted the marketing approval for the treatment of metastatic renal carcinoma patients after failure of immunotherapy.

A phase II trial (A6181040 study) on non-small cell lung cancer patients treated with sunitinib alone showed anti-tumor activity. In 63 enrolled patients treated with 4/2 schedule (4 weeks treatment, then two weeks interruption), 7 patients are confirmed partial response (overall response rate, 11%), and median progress-free time is 14.3 weeks. Presently, a phase III study is underway on non-small cell lung cancer patients followed by and now is under recruiting.

Non-small cell lung cancer cells often over-express vascular endothelial growth factor (VEGF) receptors. Besides, the expression of the VEGF ligands is also correlated with increased tumor angiogenesis, as well as shortened survival time. One study treated with VEGF-directed monoclonal antibody (bevacizumab) and VEGFR and platelet-derived growth factor receptor (PDGFR) small molecule inhibitors (sunitinib) showed that some non-small cell lung cancer patients are with anti-tumor activity.

The chemotherapy drugs, such as docetaxel and platinum-based compounds, were with evidence that they have direct cytotoxicity to cancer cells. Therefore, the investigators are paying attention to the efficacy of combining sunitinib and conventional chemotherapy in this study.

The study is designed as first line of salvage therapy on metastatic or unresectable non-small cell lung cancer patients. The main goals of this study is to evaluate the overall response rate (ORR) and duration of response (DR) of sunitinib in combinational with docetaxel and cisplatin in chemotherapy-naive advanced or metastatic non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Study Design This is a single-center, open-label, phase II clinical trial. Simon two-stage analysis is adopted.The sample size in the first stage is 16 patients. The length of study is approximately 24 months. The targeted subject is patient with metastatic or unresectable non-small cell lung cancer.

Study Endpoints Primary Endpoint Assess the response rate of sunitinib, docetaxel and cisplatin in the treatment of naïve chemotherapy metastatic or unresectable non-small cell lung cancer patients.

Secondary Endpoint

1. Time to disease progression (defined as the time period from the start of investigated medication to investigator assessed disease progression) at the end of study.
2. Duration of survival (defined as the time period from the start of investigated medication to death).
3. Safety profile of sunitinib in combination with docetaxel and cisplatin: cardiac toxicity assessed in accordance with National Cancer Institute Common Toxicity Criteria (version 3.0). The incidence of serious adverse events related to the treatment and the incidence of specific adverse events (serious and non-serious) such as gastro-intestinal perforation, wound healing complication, bleeding, hypertension, arterial thromboembolic events and proteinuria will be investigated. NCI-CTCAE criteria (version 3.0) will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female,18 years of age or older.
2. Chemotherapy-naive patients with metastatic or unresectable non-small cell lung cancer.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
4. Normal left ventricular ejection fraction (LVEF).
5. At least one unidimensionally measurable lesion with a diameter > 10 mm using CT scan.
6. Life expectancy greater than 3 months.
7. Neutrophils 1,500/L, Platelets 100,000/L, AST/ALT 2.5 ULN (< 5 ULN if liver metastases), Alkaline phosphatase 2.5 ULN, Serum bilirubin 1.5 ULN, Serum Creatinine 1.5 ULN.
8. Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate 1g of protein/24 hr.
9. Patients in this study should avoid having child. Women of childbearing potential must have a negative serum pregnancy test done 1 week prior to the administration of the study drug. She and her partner should prevent pregnancy (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) up to at least 6 months after last treatment completion or the last drug dose, whatever happens first.
10. Signed written informed consent according to ICH/GCP and the local regulations (approved by the Institutional Review Board [IRB]/Independent Ethics Committee [IEC]) will be obtained prior to any study specific screening procedures.
11. Patient must be able to comply with the protocol.

Exclusion Criteria:

1. Poor condition and inappropriate situation to enter this study, which could be determined by the principle investigator or in-charge attending physician.
2. Uncontrolled hypertension (systolic blood pressure > 160 mm Hg, diastolic blood pressure > 90 mm Hg).
3. Prior exposure to VEGF inhibitors.
4. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 0 (Patients must have recovered from any major surgery), or anticipation of need for major surgical procedure during the course of the study.
5. Planned radiotherapy for underlying disease (prior completed radiotherapy treatment allowed).
6. Clinical or radiological evidence of CNS metastases.
7. Serious non-healing wound or ulcer.
8. Evidence of bleeding diathesis or coagulopathy.
9. Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤ 6 months), myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication. Stroke in the preceding six months.
10. Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes i.e. except for anticoagulation for maintenance of potency of permanent indwelling IV catheters.
11. Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complications.
12. Ongoing treatment with large dose aspirin (> 325 mg/day) or other medications known to predispose to gastrointestinal ulceration (Continuous using NSAIDs).
13. Pregnancy (positive serum pregnancy test) and lactation.
14. Any other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
response rate by RECIST criteria | every 3 months

SECONDARY OUTCOMES:
Time to disease progression at the end of study | monthly
Duration of survival | monthly
Safety profile: cardiac toxicity assessed in accordance with National Cancer Institute Common Toxicity Criteria. NCI-CTCAE criteria (version 3.0) will be used. | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Jeng Tai, M.D., Principal Investigator — Section of Hematology-Oncology, Department of Medicine, Taipei Medical University Hospital
Locations (1):
- Section of Hematology, Department of Medicine,Taipei Medical University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Socinski MA. Adjuvant therapy of resected non-small-cell lung cancer. Clin Lung Cancer. 2004 Nov;6(3):162-9. doi: 10.3816/CLC.2004.n.029. PMID 15555217
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Mendel DB, Laird AD, Xin X, Louie SG, Christensen JG, Li G, Schreck RE, Abrams TJ, Ngai TJ, Lee LB, Murray LJ, Carver J, Chan E, Moss KG, Haznedar JO, Sukbuntherng J, Blake RA, Sun L, Tang C, Miller T, Shirazian S, McMahon G, Cherrington JM. In vivo antitumor activity of SU11248, a novel tyrosine kinase inhibitor targeting vascular endothelial growth factor and platelet-derived growth factor receptors: determination of a pharmacokinetic/pharmacodynamic relationship. Clin Cancer Res. 2003 Jan;9(1):327-37. PMID 12538485
- [Background] Papaetis GS, Syrigos KN. Sunitinib: a multitargeted receptor tyrosine kinase inhibitor in the era of molecular cancer therapies. BioDrugs. 2009;23(6):377-89. doi: 10.2165/11318860-000000000-00000. PMID 19894779
- [Background] Swanton C, Burrell RA. Advances in personalized therapeutics in non-small cell lung cancer: 4q12 amplification, PDGFRA oncogene addiction and sunitinib sensitivity. Cancer Biol Ther. 2009 Nov;8(21):2051-3. doi: 10.4161/cbt.8.21.9886. No abstract available. PMID 19816149
- [Background] Novello S, Scagliotti GV, Rosell R, Socinski MA, Brahmer J, Atkins J, Pallares C, Burgess R, Tye L, Selaru P, Wang E, Chao R, Govindan R. Phase II study of continuous daily sunitinib dosing in patients with previously treated advanced non-small cell lung cancer. Br J Cancer. 2009 Nov 3;101(9):1543-8. doi: 10.1038/sj.bjc.6605346. Epub 2009 Oct 13. PMID 19826424
- [Background] Pallis AG, Serfass L, Dziadziusko R, van Meerbeeck JP, Fennell D, Lacombe D, Welch J, Gridelli C. Targeted therapies in the treatment of advanced/metastatic NSCLC. Eur J Cancer. 2009 Sep;45(14):2473-87. doi: 10.1016/j.ejca.2009.06.005. PMID 19596191